CLINICAL TRIAL: NCT07041190
Title: PIPELINE-RSV International Trial. Pregnancy and Infant PrEparedness pLatform IN Europe (PIPELINE)- RSV International Immunisation Adaptive Platform Trial.
Brief Title: Pregnancy and Infant PrEparedness pLatform IN Europe, RSV-International Adaptive Platform Trial to Evaluate Two Approved Prevention Options to Prevent Respiratory Syncytial Virus in Infants: Maternal Vaccine to Women in Pregnancy and Monoclonal Antibody to the Infants, Given Alone or in Combination.
Acronym: PIPELINE-RSV
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: PENTA Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PIPELINE RSV-International; 2025-522194-11-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: RSV Immunization
Keywords: Pregnancy RSV Immunization; Infant RSV Immunization
MeSH Terms: interventions — abrysvo; nirsevimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Seasonal RSV monoclonal antibody (Active Comparator): RSV monoclonal antibody administered to infants at birth (or up to 7 days later) if the infant is born during the RSV season.
  Interventions: Drug: Nirsevimab
- RSV Maternal Vaccine (Active Comparator): RSV Maternal Vaccine administered to the woman in pregnancy, between 24 (or as per country guidance) and 36+6 gestational weeks.
  Interventions: Drug: Abrysvo
- RSV Maternal Vaccine + RSV infant monoclonal antibody at 4months of age (Experimental): RSV Maternal Vaccine administered to the woman in pregnancy, between 24 (or as per country guidance) and 36+6 gestational weeks, combined with infant RSV monoclonal antibody administered to the infant at 4 months of age.
  Interventions: Drug: Abrysvo; Drug: Nirsevimab

INTERVENTIONS:
Drug: Abrysvo — Maternal RSV Vaccine (MV). RSV bivalent recombinant vaccine with subgroup A and B stabilised prefusion F antigens, single intramuscular injection of 0.5 mL, administered once, in pregnancy.
  Arms: RSV Maternal Vaccine; RSV Maternal Vaccine + RSV infant monoclonal antibody at 4months of age
Drug: Nirsevimab — Infant RSV monoclonal antibody (mAb). For infants <5kg: 50mg (0.5mL in pre-filled syringe), for infants ≥5kg: 100mg (1mL in pre-filled syringe), administered as a single intramuscular injection.
  Arms: RSV Maternal Vaccine + RSV infant monoclonal antibody at 4months of age; Seasonal RSV monoclonal antibody

SUMMARY:
RSV (which stands for Respiratory Syncytial Virus) is an infection that causes cold-like symptoms and is most common during winter months. Most people with RSV infection get better by themselves but babies and younger children can become very poorly. About 1 in 15 infants with confirmed RSV within the first 12 months of life will be hospitalised, and a very small proportion will be seriously ill and may die.

Currently there are two different prevention options that can be used to prevent RSV infection in babies. One is a vaccine given to the mother during pregnancy, and the other is a monoclonal antibody given by injection to the baby. Although both prevention options work well on their own and are safe, neither provides 100% protection to the infant. It is not known whether giving both medicines, one to the mother in pregnancy and one to the infant, would provide better protection than giving only one medicine - this is what the PIPELINE-RSV study will look at.

PIPELINE-RSV-International will recruit about 1500 pregnant women from across Europe in UK, Switzerland, the Netherlands and Belgium. A parallel trial, PIPELINE-RSV-France, running in France will recruit about 1000 pregnant women in France; the protocols will align on key aspects and the data will be analysed together. The study will include three study groups with different prevention options used in each: (1) a vaccine given to the mother in pregnancy, (2) an injection given to the baby at the beginning of RSV season, or (3) both a vaccine given to the mother in pregnancy and an injection given to the baby at around 4 months of age. Each mother-baby pair will be randomly allocated to group by a computer. The numbers of babies in each of these groups who acquire RSV will be compared. In some countries only two of the three study groups may be available.

Pregnant women and their babies will be followed until the baby reaches 12 months of age. Information will be collected about medically-important side effects either the mother or the baby had from their medicine(s) and any symptoms of RSV the baby had. Visits with the mother and baby will occur at birth, and 4 and 12 months later; these will ideally be in-person at birth and at 12 months. The mother will complete questionnaires via a Web-based platform to report any non-routine in-person visits, once in pregnancy and after the baby is born twice a month or monthly (more often in the winter), to also report baby's symptoms, to report their trial experience when the baby is 4 and 12 months' old, and to provide their views on vaccination at birth, and when the baby is 4 and 12 months' old. If the baby develops symptoms that might be RSV, their mother or another caregiver will be asked to take a sample using a swab from the baby's nose or mouth, and to send it by post for testing to find out if the baby has RSV.

As well as the main research study, there are also some substudies. A questionnaire will be given to women who consent to take part, to find out their motivations for joining the study and how they prefer to receive information about taking part in studies. A small number of women will be asked to take part in a study to look at how mothers' and babies' immune systems respond to the two different study prevention options , and to investigate different ways of collecting samples from their babies. In addition, researchers will use data from the study to see whether giving both medicines is cost-effective compared with giving just one medicine.

The study might be adapted in the future to look at other medicines for preventing RSV infection, when they become available.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women

  * Pregnant woman #
  * Provide informed consent prior to study enrolment
  * Willing and able (in the Site Investigator's opinion) to comply with all study requirements
  * Above the national legal age of consent
  * Between 24+0 (or later as per national guidance) and 36+6 weeks gestation
  * Able to read and complete the eHealth questionnaire in a language in which it is available
  * Willing to receive MV in pregnancy, if allocated
  * Willing for the baby to receive infant mAb, if allocated

Infant

* Informed consent provided by the mother, and other infant legal representative (partner / co-parent) or legal guardian(s) if required by local regulations
* Live-birth to mother enrolled in the study

  * Inclusive of pregnant person of any/no gender

Exclusion Criteria:

Pregnant women

* Major illness of the maternal participant or condition of the foetus that in the opinion of the Site Investigator would substantially increase the risk associated with the woman's participation in and completion of the study
* Any suspected or confirmed condition in the foetus that in the opinion of the Site Investigator would contraindicate participation of the infant in the study
* High risk of prematurity as judged by treating clinician
* Multiple pregnancy (i.e. twins, triplets or more)
* Previous participation in the PIPELINE-RSV trial
* Receipt of any previous RSV prevention product in this pregnancy or currently participating in another interventional RSV prevention trial
* Any contraindication for receipt of intramuscular injection (bleeding diathesis or a condition associated with prolonged bleeding) or of vaccine (history of severe allergic reaction, e.g., anaphylaxis, to any component of the vaccine)
* History of Guillain Barre Syndrome

Note, all live born infants to mothers participating in the study will be included (with consent as required), but infant mAb will not be given if contraindicated.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Symptomatic RSV respiratory tract infection (RTI) in an infant, confirmed by an approved positive RSV test, by 12 months of age. | From birth to when the infant is 12 months of age.